CLINICAL TRIAL: NCT07329127
Title: Osmophobia Is Likely the Best Phenotypic Indicator of Migraine: A Prospective, Non-Interventional, 6-Month Longitudinal Study
Brief Title: The Prevalence of Osmophobia in Migraine and Tension-Type Headache Patients and Its Association With Migraine Symptoms Over a Period of 6 Months
Status: Completed | Type: Observational
Sponsor: National and Kapodistrian University of Athens (Other)
Responsible Party: Principal Investigator, Sofia Tsanoula, Neurology Resident, Neurology Department of Hôpitaux Universitaires de Genève, PHD Student, National and Kapodistrian University of Athens
Other Study IDs: ΨΤΧ446Ψ8Ν2-4Β5
Record Dates: First submitted 2025-12-04; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-12

CONDITIONS: Migraine; Tension Headache
Keywords: migraine; osmophobia; Predictive markers; sensory hypersensitivity; diagnostic criteria
MeSH Terms: conditions — Migraine Disorders; Tension-Type Headache

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients with episodic or chronic migraine with or without aura
- Patients with episodic or chronic tension type headache

SUMMARY:
The goal of this observational study is to learn about the frequency and diagnostic value of osmophobia, which is a sensitivity to smell, in people with migraine compared to those with tension-type headache. The main question it aims to answer is:

Does osmophobia reliably indicate a migraine rather than a tension-type headache?

Participants diagnosed with migraine or tension-type headache at the Headache Outpatient Department of Aeginition Hospital of Athens will record their headaches and any sensitivity to smells using a headache diary and a special osmophobia calendar over a period of six months. They will also complete questionnaires about migraine burden and related health conditions.

DETAILED DESCRIPTION:
Main research question and why it is important:

Our aim is to estimate the frequency of osmophobia in migraine and tension-type headache. The significance of the result lies in the possible use of osmophobia as a diagnostic tool in the diagnostic criteria for migraine.

-Main Report (based on the above main research question): This is a prospective, non-interventional, six-month longitudinal study in which patients visiting the headache clinic will undergo a special semi-structured interview specific to headaches, in accordance with the electronic program of the Greek Headache Society (individual, family, frequency and duration of attacks, intensity of pain), which includes the MIDAS (Migraine Disability Assessment) and HIT-6(Headache Impact Test) scales. They will be given a special headache diary and a special diary for osmophobia, which they will complete and reassess over a period of 6 months.

-Study tools: Headache diary, Specialised osmophobia diary, MIDAS(Migraine Disability Assessment), HIT-6(Headache Impact Test), BECK depression scale, Written consent form

The migraine diary includes specific information about the nature of each attack (duration, intensity, presence of aura, worsening with activity) and the presence of accompanying symptoms (nausea, vomiting, photophobia, phonophobia), while the osmophobia diary specifies the characteristics of osmophobia (intensity, duration, temporal correlation with headache, type of odors, whether or not odors cause headache). The MIDAS and HIT-6 scales determine quality of life in migraine, and the BECK scale determines mood status.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a diagnosis of migraine or tension-type headache (ICHD-3)
2. Age >16 years
3. Patients with or without medication overuse headache
4. Patients with or without prophylaxis
5. Patients with or without comorbidity with mood disorders
6. Patients will have signed informed consent to participate in the study

Exclusion Criteria:

1. Patients with primary or secondary anosmia
2. Inability to obtain written consent

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients visiting the Headache Outpatient Department of Eginition Hospital of Athens
Sampling Method: Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2024-01-08 (Actual); Primary Completion 2024-12-30 (Actual); Study Completion 2024-12-30 (Actual)

PRIMARY OUTCOMES:
The frequency of osmophobia in migraine and tension-type headache | At baseline assessment over a six month period
  Our aim is to estimate the prevalence of osmophobia in migraine and tension type headache in order to clarify its significance as a diagnostic tool for migraine

SECONDARY OUTCOMES:
The correlation of osmophobia with headache type and symptoms and the calculation of its sensitivity and specificity | At baseline assessment over a six month period
  Our secondary aim is to estimate the correlation of osmophobia with the type and characteristics of migraine and tension-type headache, e.g. with accompanying symptoms such as nausea or vomiting, but also with comorbidities such as depression disorders. In addition, the sensitivity and specificity of osmophobia as a diagnostic criterion for migraine, as well as the sensitivity, specificity, positive and negative predictive values will be calculated for each different accompanying symptom of migraine.

CONTACTS AND LOCATIONS:
Locations (1):
- Aeginition Hospital of Athens, Athens, Greece

IPD SHARING:
Plan to Share IPD: Undecided